CLINICAL TRIAL: NCT06447285
Title: Early, Objective Detection of Autism.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SensoDetect (Industry)
Collaborators: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: HA-01-R-104
Record Dates: First submitted 2024-05-19; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder
Keywords: ABR (Auditory brainstem response)
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autism spectrum disorders group (Active Comparator): All patients shall be diagnosed according to ADOS15 and DSM-517 criteria by an experienced physician. ADOS is a diagnostic tool considered the "gold standard" in ASD diagnostics.18,19 The children with confirmed diagnoses of autism will be assessed by a senior psychologist using the Stanford-Binet Intelligence Scales - Fifth edition (SB-5)21 to ensure that all ASD patients have an IQ of 70 or above. ASD patients with lower IQ will form a distinct group for specific evaluation.
  Using sensodetect BERA technology we will in the present study pay attention to wave I-VII amplitude as well as latencies and interpeak intervals to broaden the perspective and allow a better comparison of both groups.
  Group differences between autistic and TD groups will be tested intra-individually and between groups and presented.
  Interventions: Diagnostic Test: SensoDetect BERA technology
- totally developed group (Active Comparator): All patients shall be diagnosed according to ADOS15 and DSM-517 criteria by an experienced physician. ADOS is a diagnostic tool considered the "gold standard" in ASD diagnostics.18,19 The children with confirmed diagnoses of autism will be assessed by a senior psychologist using the Stanford-Binet Intelligence Scales - Fifth edition (SB-5)21 to ensure that all ASD patients have an IQ of 70 or above. ASD patients with lower IQ will form a distinct group for specific evaluation.
  Using sensodetect BERA technology we will in the present study pay attention to wave I-VII amplitude as well as latencies and interpeak intervals to broaden the perspective and allow a better comparison of both groups.
  Group differences between autistic and TD groups will be tested intra-individually and between groups and presented.
  Interventions: Diagnostic Test: SensoDetect BERA technology

INTERVENTIONS:
Diagnostic Test: SensoDetect BERA technology — All recruited participants are to be tested using SensoDetect's patented technology. All tests shall be performed in a quiet and darkened room. Participants will be asked to be comfortably seated in an armchair in a resting position (part 1 only). Surface electrodes will then be attached to the skin over the mastoid bones behind the left and right ear, with a ground electrode on one arm. Two reference electrodes will also be placed on the forehead. Before each test session, the procedure shall be fully explained to the test subject or parents.
  The subjects will then be instructed to relax with their eyes closed and are permitted to fall asleep (with modifications in part 3). The test will require no active participation other than being subjected to sound stimulation. The subjects will be tested one at a time, and the duration of the testing procedure will be 15 min.

SUMMARY:
1- To test the hypothesis that using the SensoDetect Brainstem Evoked Response Audiometry (BERA) technology may be an effective support tool for pediatricians to detect autism.

DETAILED DESCRIPTION:
This study will be conducted through two phases:

Phase I: A case-control study.

This will be done at Princess Noura University/ King Abdullah Abdulaziz University Hospital, Riyadh, Kingdom of Saudi Arabia from January 2024 to January 2027.

The SensoDetect BERA technology previously described8,9,13,14 will be used in all parts of the study in the following way:

All recruited participants are to be tested using SensoDetect's patented technology. All tests shall be performed in a quiet and darkened room. Participants will be asked to comfortably sit in an armchair in a resting position (part 1 only). Surface electrodes will then be attached to the skin over the mastoid bones behind the left and right ear, with a ground electrode on one arm. Two reference electrodes will also be placed on the forehead. Before each test session, the procedure shall be fully explained to the test subject or parents.

The subjects will then be instructed to relax with their eyes closed and are permitted to fall asleep (with modifications in part 3). The test will require no active participation other than sound stimulation. The subjects will be tested one at a time, and the duration of the testing procedure will be 15 min.

The method is based on an electrophysiological test battery that emits 1024 click sounds divided into 4 sessions for 14 minutes. The data analysis software uses advanced mathematical algorithms and Artificial intelligence (AI) to analyze and distinguish the patient's markers and compare them with diagnostic and non-diagnostic groups. BERA is CE and MDD (MDD stands for Medical Device Directive and is an approval for the device to be used under European law) approved. SensoDetect holds the ISO standard under medical technical products 13485:2016. After the test is completed, the result will be sent for analysis using SensoDetect's analytical software (SensoLytics). The AI classification model used for analyzing traits and predicting diagnosis is Gaussian Naïve Bayes.

ELIGIBILITY:
Phase I:

Inclusion Criteria:

- All patients attending the clinic of Autism.

Exclusion Criteria:

* Hearing impairment
* Down syndrome
* Cerebral Palsy
* Significant brain damage Intellectual disability.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2024-05-29 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
wave I-VII amplitude | phase 1 of this study one year
  Wave I-VII amplitude allow comparison of both groups. Group differences between autistic and totally developed (TD) groups will be tested intra-individually and between groups and presented.
Wave I-VII latencies | phase 1 of this study one year
  wave I-VII latencies to broaden the perspective and allow a better comparison of both groups.
  Group differences between autistic and TD groups will be tested intra-individually and between groups and presented.
Wave I-VII interpeak intervals | phase 1 of this study one year
  Wave I-VII interpeak intervals allow a comparison of both groups. Group differences between autistic and TD groups will be tested intra-individually and between groups and presented.

IPD SHARING:
Plan to Share IPD: No